CLINICAL TRIAL: NCT05312567
Title: Randomized, Double-Blind, Plac.-Controlled Clinical Study to Compare the Efficacy of FP-101 60mg b.i.d. vs. Placebo for the Treatment of Moderate-to-Severe Hot Flashes in Peri- and Post-menopausal Women Over a Period of 1-Week.
Brief Title: FP-101 Versus Placebo in the Treatment of Menopausal Vasomotor Symptoms
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Fervent Pharmaceuticals (Industry)
Collaborators: ICON plc (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 2021-FERV
Record Dates: First submitted 2022-03-28; First posted 2022-04-05 (Actual); Last update posted 2023-10-26 (Actual); Status verified 2023-10

CONDITIONS: Vasomotor Symptoms; Menopause

STUDY DESIGN:
Intervention Model Description: Randomized, double-blind, parallel-group, placebo-controlled study to compare patient-reported changes in VMS for the IMP vs. placebo. The study will be run as a fully decentralized clinical trial.
Who Masked: Participant, Investigator
Masking Description: Matching placebo tablets. Double-blind treatment packaging and dispensation.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Active Treatment (FP-101) (Experimental): White to off-white extended-release, round tablets containing FP-101.
  Interventions: Drug: FP-101
- Matching placebo (Placebo Comparator): White to off-white round tablets without the active ingredient but otherwise matching in size and appearance.
  Interventions: Drug: FP-101

INTERVENTIONS:
Drug: FP-101 — daily oral tablet administration (b.i.d.)

SUMMARY:
This Phase II proof of concept study is designed to assess the safety and efficacy of FP-101 (60mg b.i.d.), an extended-release oral tablet product, compared to a matching placebo in the treatment of moderate-to-severe hot flashes in peri- and post-menopausal women over a period of 1-week.

DETAILED DESCRIPTION:
This randomized, double-blind, parallel-group, placebo-controlled, clinical trial is designed to compare patient-reported changes in Vasomotor Symptoms (VMS) for FP-101 vs. placebo in peri- and post-menopausal women. The study will be run as a fully decentralized clinical trial (DCT), by use of components such as electronic Consent (eConsent), mobile/tele health visits, electronic Patient Reported Outcomes (ePROs), and direct-to-participant shipping of the (investigational medicinal product (IMP). The DCT approach to this study will rely on a digital platform through which subjects can consent, enroll, and interact with the PI and study staff. Proper regulatory framework and technology use will ensure compliance with Good Clinical Practice (GCP), ethics & legal/regulatory requirements.

Healthy peri- and post-menopausal women (>45 years of age) suffering from VMS will be recruited if they have >=7- 8 moderate to severe hot flushes per day at baseline. After meeting all eligibility criteria subjects will be enrolled and start a 1-week run-in period to identify/eliminate placebo responders, as well as to exclude subjects who have difficulty completing the eDiary. Any Adverse Events (AEs) during the run-in period will serve as baseline for the safety assessments at the end of the treatment period.

Eligible subjects will undergo a tele health baseline visit during which the criteria for inclusion in the treatment period will be confirmed. Over a 1-week treatment period, subjects will complete a daily electronic Diary (eDiary) to record any AEs and the frequency and severity of hot flashes during the past 12hr interval. In the morning, subjects will record the number of awakenings during the past night and the number of night sweats.

The PI will conduct an end-of-study visit with each of the subjects randomized to the study medications to review safety and efficacy data, complete a Patient Global Improvement Scale, and clarify any open issues with the subjects.

------------------------------

ELIGIBILITY:
Inclusion Criteria:

* Peri- and Post-Menopausal female subjects (>45 yrs) experiencing a min of 7-8 moderate to severe hot flashes per day
* Able/willing to provide informed consent.
* Able/willing to complete all study procedures and visits.
* Able/willing to not use any over-the-counter (OTC) cough & cold medications that contain the IMP active during the study.

Exclusion Criteria:

* Subject exhibits positive home pregnancy test at screening or any time during study
* Subject currently taking any form of Hormone Therapy (HT), including local estrogen therapies
* Subject currently taking tamoxifen, other selective estrogen receptor modulators, or other hormone deprivation therapy.
* Subject with history of serotonergic syndrome
* Subject is currently taking monoamine oxidase inhibitors (MAOIs) (or for 2 weeks after stopping the MAOI drug), antidepressants, thioridazine, pimozide, cannabidiol, opioids, antipsychotic agents, antiretroviral agents, quinidine, quinine, or other medications for VMS such as Brisdelle® (paroxetine mesylate), clonidine and gabapentin.
* Subject is currently taking a dietary/herbal supplement(s) to manage VMS, such as soy isoflavones or black cohosh.
* Subject has uncontrolled diabetes, a history of hypertension & is not on a stable dose of antihypertensive medications for at least 30 days prior to screening.
* Subject has clinically unstable cardiac disease, including atrial fibrillation, symptomatic brady- or tachy-arrhythmias, congestive heart failure (NYHA class II, III, and IV), or symptomatic atherosclerotic cardiovascular disease (coronary artery disease, carotid artery disease or peripheral artery disease) or history of myocardial infarction or stroke within 2 years of enrolment in the study.
* Subject reports medical history suggestive of impaired liver/kidney function or, in the PI's opinion, exhibits liver/kidney function impairment to the extent that the subject should not participate in the study.
* Subject has biliary tract disease, adrenal cortical insufficiency, or any other medical condition that, in the PI's opinion (and after discussion with the medical monitor), is considered inadequately treated and precludes entry into the study.
* Subject has thyroid disease, unless subject is clinically stable with normal thyroid indices and is on maintenance thyroid medication (e.g., levothyroxine or liothyronine) for ≥6 months prior to screening.
* Subject has a history of, or is currently presenting with, substance use disorder as defined by the 5th Edition of the Diagnostic and Statistical Manual of Mental Disorders (DSM). Subject has a history of psychiatric disorders, including a lifetime history of major depressive disorder, bipolar disorder, panic disorder, generalized anxiety, psychotic disorders, suicidality or suicidal ideation, or post-traumatic stress disorder.
* Subject is currently participating in another clinical trial
* Subjects who were determined to be placebo responders or non-compliant during the 1-week run-in period.

Min Age: 46 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes — Peri- and Post-menopausal women
Enrollment: 105 (Actual)
Dates: Start 2021-03-24 (Actual); Primary Completion 2023-04-05 (Actual); Study Completion 2023-07-31 (Actual)

PRIMARY OUTCOMES:
Change in the frequency (average daily number) of moderate-to-severe hot flashes. | Recorded every 12 hrs over a 1-week treatment period.
  Subjects use a digital platform to record hot flash frequency in a daily eDiary.

SECONDARY OUTCOMES:
Change in the severity (average daily rating) of moderate-to-severe hot flashes. | Recorded every 12 hrs over a 1-week treatment period.
  Subjects use digital platform to record hot flash severity (3-point scale) in a daily eDiary.
Change in nighttime awakenings (average daily number) with or without night sweats. | Recorded every morning over a 1-week treatment period.
  Subjects use daily eDiary to record nighttime awakenings & night sweats frequency.
Evaluate the clinical meaningfulness of VMS changes after 1-week of treatment. | After 1 week of treatment at the end-of-study visit.
  Completing validated Patient Global Improvement Scale (7-point) with PI.

OTHER OUTCOMES:
Any Adverse Events and Concomitant Medications | Recorded as needed/every 12 hrs over a 1-week treatment period.
  Subjects will use daily eDiary to record any AEs and concomitant medications

CONTACTS AND LOCATIONS:
Overall Officials: Helmut H Albrecht, MD, Study Director — Lumanity
Locations (12):
- United States (12):
  - Torrance Clinical Research Institute, Lomita, California
  - Long Beach Clinical Trial Services, Long Beach, California
  - Provideré Research Inc., West Covina, California
  - Inpatient Research Clinic, Hialeah, Florida
  - The Angel Medical Research Corporation, Miami Lakes, Florida
  - Suncoast Clinical Research - Pasco County, New Port Richey, Florida
  - Cary Medical Group, Cary, North Carolina
  - Raleigh Medical Group, Raleigh, North Carolina
  - Clinical Research of Philadelphia, Philadelphia, Pennsylvania
  - Coastal Carolina Research Center, North Charleston, South Carolina
  - ICON Early Phase Services, San Antonio, Texas
  - Discovery Clinical Trials - Stone Oak, San Antonio, Texas

IPD SHARING:
Plan to Share IPD: No
No plans to share data with other researchers